CLINICAL TRIAL: NCT04960267
Title: Use of Pre-peritoneal Drainage in rTAPP - a Comparative Study With Laparoscopic TEP
Brief Title: Use of Pre-peritoneal Drainage in rTAPP - a Comparative Study
Acronym: DrainrTAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Joe King-Man Fan, Consultant, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERN-rTAPPDRAIN-01
Record Dates: First submitted 2021-06-10; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hernia, Inguinal
Keywords: hernia; inguinal; seroma; drain; robotic; TAPP; rTAPP
MeSH Terms: conditions — Hernia, Inguinal; Hernia; Seroma

STUDY DESIGN:
Intervention Model Description: The safety and efficacy of pre-peritoneal drain after TEP has been validated in our previous studies - which can effectively reduce seroma formation post-operatively and safe in clinical use. We shall extend the indication of pre-peritoneal drainage after robotic TAPP, results will be compared with our retrospective cohort from previous studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Use of pre-peritoneal drainage after rTAPP (Experimental): Use of pre-peritoneal drainage after rTAPP
  Outcomes will be compared with retrospective cohort from our previous experiments
  Interventions: Device: Use of pre-peritoneal drainage after rTAPP

INTERVENTIONS:
Device: Use of pre-peritoneal drainage after rTAPP — Use of pre-peritoneal drainage after rTAPP

SUMMARY:
The safety and efficacy of pre-peritoneal drain after TEP has been validated in our previous studies - which can effectively reduce seroma formation post-operatively and safe in clinical use. We shall extend the indication of pre-peritoneal drainage after robotic TAPP, results will be compared with our retrospective cohort from previous studies.

DETAILED DESCRIPTION:
The safety and efficacy of pre-peritoneal drain after TEP has been validated in our previous studies - which can effectively reduce seroma formation post-operatively and safe in clinical use. We shall extend the indication of pre-peritoneal drainage after robotic TAPP, results will be compared with our retrospective cohort from previous studies.

Criteria of enrolling into trial is same as our previous experiment: aged 18-80, unilateral, first occurrence, reducible, non-inguino-scrotal inguinal hernia fit for GA for minimally invasive hernia repair. Routine robotic TAPP performed in standardized manner and pre-peritoneal drains are placed for drainage of 23 hours post-operatively. Drain output, pain scores, status of seroma formation (clinical, USG detected), post-operative recovery and recurrence will be monitored and compared.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral,
* First occurrence
* Reducible inguinal hernia

Exclusion Criteria:

* Not fit for GA,
* Bilateral hernia
* Recurrent hernia
* Irreducible hernia
* Inguino-scrotal extension hernia
* Non-inguinal hernia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Pre-peritoneal Drainage output after rTAPP | at 23 hours post-operation
  Pre-peritoneal Drainage output (ml) after rTAPP

SECONDARY OUTCOMES:
Seroma formation | day 7, 1 month
  Clinical detectable seroma and size of seroma detected by USG after rTAPP with pre-peritoneal drainage

CONTACTS AND LOCATIONS:
Overall Officials: Joe KM FAN, MBBS MS, Principal Investigator — The University of Hong Kong-Shenzhen Hospital
Locations (1):
- Department of Surgery, The University of Hong Kong - Shenzhen Hospital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan JKM, Liu J, Chen K, Yang X, Xu X, Choi HK, Chan FSY, Chiu KWH, Lo CM. Preperitoneal closed-system suction drainage after totally extraperitoneal hernioplasty in the prevention of early seroma formation: a prospective double-blind randomised controlled trial. Hernia. 2018 Jun;22(3):455-465. doi: 10.1007/s10029-018-1731-2. Epub 2018 Jan 13. PMID 29332240
- [Background] Li J, Zhang W. Comment to: Preperitoneal closed-system suction drainage after totally extraperitoneal hernioplasty in the prevention of early seroma formation: a prospective double-blind randomised controlled trial. Fan JKM, Liu J, Chen K, Yang X, Xu X, Choi HK, Chan FSY, Chiu KWH, Lo CM. Hernia. 2018 Jun;22(3):467-468. doi: 10.1007/s10029-018-1762-8. Epub 2018 Apr 21. No abstract available. PMID 29681017
- [Background] Fan JKM, Liu J, Chen K, Yang X, Xu X, Choi HK, Chan FSY, Chiu KWH, Lo CM. Reply to Comment to: Preperitoneal closed-system suction drainage after totally extraperitoneal hernioplasty in the prevention of early seroma formation: a prospective double-blind randomized controlled trial. Hernia. 2018 Jun;22(3):469-470. doi: 10.1007/s10029-018-1764-6. Epub 2018 Apr 21. No abstract available. PMID 29681018
- [Background] Gao D, Wei S, Zhai C, Chen J, Li M, Gu C, Wu H. Clinical research of preperitoneal drainage after endoscopic totally extraperitoneal inguinal hernia repair. Hernia. 2015 Oct;19(5):789-94. doi: 10.1007/s10029-014-1310-0. Epub 2014 Sep 20. PMID 25238803
- [Background] Fan JKM, Yip J, Foo DCC, Lo OSH, Law WL. Randomized trial comparing self gripping semi re-absorbable mesh (PROGRIP) with polypropylene mesh in open inguinal hernioplasty: the 6 years result. Hernia. 2017 Feb;21(1):9-16. doi: 10.1007/s10029-016-1545-z. Epub 2016 Nov 26. PMID 27889845
- [Result] Liu JW, Chen KJ, Xu XH, Deng Y, Zhang H, Chan FSY, Kim HJ, Fan JKM. Does the use of monopolar energy as the preferred mode of dissection effectively reduce seroma formation in laparoscopic total extra peritoneal hernioplasty? A prospective double-blinded randomized control trial. Hernia. 2020 Aug;24(4):821-829. doi: 10.1007/s10029-020-02136-3. Epub 2020 Feb 18. PMID 32072340